CLINICAL TRIAL: NCT05990426
Title: The Impact of Alternate Day Fasting After Surgery for Patients Undergoing ChemoTherapy (FAST Study)
Brief Title: Alternate Day Fasting After Surgery for Patients Undergoing Chemotherapy
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jenna Marcus, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU00217844
Record Dates: First submitted 2023-04-14; First posted 2023-08-14 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ovary Cancer; Endometrial Cancer; Uterine Cancer
Keywords: chemotherapy; peripheral neuropathy; intermittent fasting
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Neoplasms; Peripheral Nervous System Diseases; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: This study is an unblinded two-arm randomized controlled trial to investigate the effects of alternate day fasting in ovarian and uterine cancer patients undergoing chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FAST Group (Experimental): The FAST intervention will consist of one week of alternate day fasting (ADF) using the sandwich model at the start of each cycle of chemotherapy, for a total of 6 weeks of ADF. Patients will be instructed on how and what they may consume on fasting days.
  Interventions: Behavioral: FAST Intervention
- Control Group (No Intervention): Participants in the control arm will be instructed to eat as desired throughout their entire chemotherapy treatment course. Control group participants will not receive any special study- related instructions or direction regarding food and drinks consumed during chemotherapy.

INTERVENTIONS:
Behavioral: FAST Intervention — Participants will alternate fasting days (FAST) with unrestricted eating (OFF, or "Feast") days, for one week surrounding the start of each chemotherapy cycle. The participants will fast for two consecutive days in the middle of the ADF week - the day prior to chemotherapy start date, and chemotherapy day 1 for each cycle. Participants will consume regular diet (OFF/Feast) during other days 5-18 of each cycle.
  Other Names: Alternate Days Fasting Dietary Regimen
  Arms: FAST Group

SUMMARY:
Endometrial cancer is the most common gynecologic cancer and ovarian cancer is the most lethal. The management of both advanced cancers is a combination of chemotherapy and surgery. Standard of care chemotherapeutic treatment for uterine and ovarian cancers is toxic and severely disruptive to the patient's quality of life with the potential for devastating short and long-term side effects. The role of fasting and ketogenic diets has been evaluated in a mixed cancer population and previously shown to be safe. There is no data specifically addressing the impact of a fasting diet regimen on side effects of chemotherapy during treatment for ovarian and endometrial cancers in the front-line setting. The information gathered from this study will inform future trials about the role of time-restricted eating and its impact on side-effects associated with chemotherapy as well as its role in improvement of quality of life for women afflicted with these debilitating diseases.

DETAILED DESCRIPTION:
Uterine cancer is the most common gynecologic cancer diagnosed in women and the fourth most common cancer to be diagnosed in females with an estimated 65,950 cases that will be diagnosed this year in the United States. Although not as common as endometrial cancer, ovarian cancer is the fifth most lethal cancer in females with an estimated 19,880 cases diagnosed this year. Standard of care treatments such as chemotherapy are toxic and severely disruptive to the patient's quality of life with potential short and long-term devastating side effects. The management of advanced gynecologic cancers of the uterus and ovary is often with a combination of surgery and chemotherapy in medically stable patients. The sequence of treatment is dependent on the patient's medical conditions, disease distribution and likelihood of complete resection at the time of surgery. Even when surgery results in complete resection in those with advanced disease, systemic treatment with chemotherapy is frequently prescribed. First line treatment for advanced uterine and ovarian cancer with carboplatin and paclitaxel has been shown to be tolerable and effective. However, these drugs often have a wide range of toxic side effects associated with their administration and may require treatment delays or dosing adjustments for patients to complete the prescribed treatment. In addition to hematologic toxicity and metabolic derangements, systemic chemotherapy often has debilitating side effects associated with treatment such as peripheral neuropathy. Supportive medications for side effects associated with chemotherapy are often given to patients for self-administration at home to combat symptoms in the several days following infusion, but there are limited interventions available to help patients further and with long term toxicities. New strategies are needed to help patients better tolerate these taxing side effects to improve patient outcomes and quality of life.

The effect of diet in rodents is well studied and has shown restriction of calories results in improved lifespan, and delayed onset of age associated diseases such as hypertension, diabetes, autoimmune conditions and cancer. With respect to chemotherapy administration in humans, the concept of differential stress resistance has been published and demonstrates protection of normal cells during periods of fasting where, conversely cancer cells become more susceptible to chemotherapy. This has been applied in few human studies where the impact of diet on cancer treatment was evaluated across a variety of cancer diagnoses and was found be safe and without worsening side effects from treatment. In time-restricted eating, participants eat within a specific time (eating window) and fast for the rest of the day (fasting window) every day.

There are several definitions and descriptions of intermittent fasting (IF). There are 2 components to the fasting regimen: (1) the duration of the actual time fasting (hours) and (2) the schedule of the periods of fasting (days, weeks, months). Alternate day fasting (ADF) is defined as 24-hour periods of fasting alternating with 24-hour periods of eating/feasting. This can be modified and extend the fasting window up to periods of 72 hours as previously studied in cancer populations and has been feasible and tolerable. The fasting schedule is then either prolonged over periods of weeks or short-term over a period of days. Prolonged fasting has been used for caloric restriction and long-term weight loss, which is not ideal in a cancer population. We chose this short-term, modified alternate day fasting regimen to both limit weight loss and center the prescribed "fasting window" around administration of chemotherapy when we expect to see the largest benefit in terms of reduction of toxic chemotherapy-related side effects. In addition, food intake rapidly initiates a cascade of biochemical responses to process the incoming nutrients. In contrast, during fasting, the body mobilizes stored energy. Specifically, the mechanistic target of rapamycin complexes-1 and -2 (mTORC1 and mTORC2) are regulated by nutrient availability, and loss of mTOR signaling partially mediates the cellular effects of fasting interventions on cancer cells. In muscles, caloric intake activates mTOR signaling within 30 minutes of eating to yield an anabolic state, with peak mTORC1 activity at approximately 60-90 minutes. Subsequently, mTORC1 is gradually deactivated. Approximately 12-16 hours after food absorption, a metabolic switch is activated in which the primary source of energy shifts from glucose to fat and ketones. This metabolic switch, mediated by decreased mTOR signaling, is key for prolonged fasting (>~16 hours) to be effective. Using ADF helps in initiating this metabolic switch several times before, during, and after chemotherapy and might increase the benefit of fasting. Another form of intermittent fasting is alternate-day fasting (ADF) which is defined as alternating between fasting day (0-25% of energy needs) and feasting day (eating as desired). Preliminary studies in ovarian cancer patients suggest that restricting energy and/or protein intake at the time of chemotherapy might help reduce chemotherapy-related side effects and improve patients' quality of life. Of particular concern in an ovarian cancer patient population is malnutrition and the contribution of a time restricted eating intervention on weight loss. Intermittent fasting and, more specifically, short-term fasting, has been used in several pilot studies and has shown beneficial effects among the gynecologic and breast cancer populations without weight loss or serious adverse events. There are few published studies which look at multiple cancer types in each study and evaluate patients at variable timepoints in their treatment (ie. Initial vs recurrent disease). The effect of alternate day fasting during front-line chemotherapy on chemotherapy-associated side effects and quality of life has never been tested. Here we propose a dietary strategy in gynecologic cancer patients undergoing their first line of treatment to study the impact of intermittent fasting in patients with uterine and ovarian cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Female; ≥ 18 years of age
2. Confirmed or high suspicion for endometrial, ovarian, fallopian tube or primary peritoneal cancer, and are able and expecting to undergo adjuvant chemotherapy following hysterectomy for treatment of disease, as determined by their treating physician
3. Fluent in spoken and written English
4. Own a smart phone
5. Have access to the internet to complete surveys
6. ECOG status of 0 or 1
7. Willingness to sign informed consent form

Exclusion Criteria:

1. Patients who are not planning to undergo chemotherapy at Northwestern Medicine
2. Patients engaged in shift work (i.e., those who work nights, 3rd shift)
3. BMI of 50+ or those with a diagnosed eating disorder. Patients who take medications for blood glucose regulation (e.g. insulin), and/or require treatment with therapeutic doses of anticoagulants will be excluded.
4. Patients who have been diagnosed with medication-dependent diabetes, recent myocardial infarction, stroke, pulmonary embolus, renal failure, or any condition that may preclude ability to tolerate a short-term fast will be excluded.
5. Patients who take medications where conditions may be influenced in the presence of fasting (e.g. hypertension, electrolyte abnormalities, migraines) will be monitored by their treating physician for any necessary adjustments in these medications.
6. Patients whose oncologist has not provided clearance for their participation
7. Unable or unwilling to follow a diet regimen or participate in ketone measurements
8. ECOG status greater than 1
9. Patients who have undergone prior systemic therapy to treat a malignancy in the last 2 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assessment Compliance | 18 weeks
  Assessment compliance will be defined as missing no more than 75% of indicated Biosense measurement (i.e. no more than number of cycles × 7 measurements), which roughly corresponds to no more than 1 missed measurement per day of fasting period. The study will be considered feasible in terms of assessment compliance if at least 80% of all patients are compliant.
Treatment Compliance | 18 weeks
  Treatment compliance will be defined among patients on FAST as the proportion of measurements on fasting days when the patient is in ketosis (i.e., ACE score > 5, or ketone levels of 0.5+ mmol/L). FAST treatment will be considered feasible in this patient population if >80% of patients in the FAST arm are compliant with treatment.
Fasting non-compliance | 18 weeks
  Fasting non-compliance will be defined as anyone who began fasting but was not compliant with completing the 48-hour fast. Anyone who started ADF by following low caloric (equal or less than 400 cal) fast within 24 hours of C1D1 chemo regimen will be considered fasting compliant. Patients randomized to the intervention arm will be considered evaluable if they start their fasting diet regimen within 24 hours prior to starting day 1 of their first chemotherapy cycle (C1D1) and if they fast for three out of the four 24-hour long fasting windows within each of the six chemotherapy cycles. Patients randomized to the control arm will be considered evaluable if they started chemotherapy. Fasting non-compliance will be measured by number of participants meeting the above definition.

SECONDARY OUTCOMES:
Adverse events and toxicity | 18 weeks
  Assess differences in expected toxicities associated with chemotherapy administration using Common Terminology Criteria for Adverse Events (CTCAE)
  Safety definition: we expect toxicity profile to be similar between the two arms, although formally testing the Adverse Event (AE) rates will be underpowered. After every 6 patients have been randomized (4+2 in the two arms), the PI will review cumulative toxicity data by arm. If a high proportion of patients in the AFT arm has a particular type of AE which has substantially lower prevalence or is not observed in the non-AFT arm, enrollment may be paused to further evaluate the reasons and supportive care of these unexpected AE's.
  Patients will be considered evaluable for safety if they started any of the study treatments (ADF and chemotherapy).
Neuropathic Pain | 18 weeks
  Assess differences in Patient Reported Outcomes (PROs) utilizing Patient Reported Outcomes Measurement Information System (PROMIS) surveys for neuropathic pain
Physical Function | 18 weeks
  Assess differences in Patient Reported Outcomes (PROs) utilizing Patient Reported Outcomes Measurement Information System (PROMIS) surveys for physical function

OTHER OUTCOMES:
Cancer Related Fatigue | 18 weeks
  Assess differences in Patient Reported Outcomes (PROs) utilizing Patient Reported Outcomes Measurement Information System (PROMIS) surveys for cancer related fatigue
Molecular biomarker: Insulin | 18 weeks
  Insulin concentration from human serum will be measured and reported as pg/ml using enzyme-linked immunosorbent assay (ELISA) performed by the Comprehensive Metabolic Core Facility at Northwestern University's Feinberg School of Medicine
Molecular biomarker: insulin-like growth factor-1 | 18 weeks
  Insulin-like growth factor-1 concentration from human serum will be measured and reported as pg/ml using enzyme-linked immunosorbent assay (ELISA) performed by the Comprehensive Metabolic Core Facility at Northwestern University's Feinberg School of Medicine
Molecular biomarker: Insulin-like growth factor Binding Protein-1 | 18 weeks
  Insulin-like growth factor Binding Protein-1 concentration from human serum will be measured and reported as pg/ml using enzyme-linked immunosorbent assay (ELISA) performed by the Comprehensive Metabolic Core Facility at Northwestern University's Feinberg School of Medicine
Molecular biomarker: Estrone | 18 weeks
  Estrone concentration from human serum will be measured and reported as pg/ml using enzyme-linked immunosorbent assay (ELISA) performed by the Comprehensive Metabolic Core Facility at Northwestern University's Feinberg School of Medicine
Molecular biomarker: Progesterone | 18 weeks
  Progesterone concentration from human serum will be measured and reported as pg/ml using enzyme-linked immunosorbent assay (ELISA) performed by the Comprehensive Metabolic Core Facility at Northwestern University's Feinberg School of Medicine
Molecular biomarker: Testosterone | 18 weeks
  Testosterone concentration from human serum will be measured and reported as pg/ml using enzyme-linked immunosorbent assay (ELISA) performed by the Comprehensive Metabolic Core Facility at Northwestern University's Feinberg School of Medicine
Patient Satisfaction Questionnaire | 18 weeks
  Each patient's satisfaction with the diet intervention during chemotherapy will be assessed using a 12-question survey distributed to the participants randomized to the FAST intervention group. Participants will be asked questions regarding their satisfaction, feasibility, and ease of following the diet regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Marcus, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No